CLINICAL TRIAL: NCT02051543
Title: Investigating Affective Mechanisms of Behavioral Sleep Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Erin Koffel, Psychologist, Minneapolis Veterans Affairs Medical Center
Other Study IDs: vamc-eak-1
Record Dates: First submitted 2014-01-28; First posted 2014-01-31 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brief Behavioral Treatment of Insomnia-Military Version (Experimental)
  Interventions: Behavioral: Brief Behavioral Treatment of Insomnia -Military Version

INTERVENTIONS:
Behavioral: Brief Behavioral Treatment of Insomnia -Military Version

SUMMARY:
Insomnia is a highly prevalent condition and costly national public health problem and a transdiagnostic risk factor for the development of a number of internalizing/emotional disorders, as well as associated functional impairment. Interestingly, sleep treatments appear to reduce anxiety and depression in addition to improving sleep. Given the substantial individual and societal costs of insomnia and associated mental illness, there is an urgent need to better understand the mechanism through which sleep treatments improve daytime symptoms of depression and anxiety in order to enhance the efficacy of sleep treatments and ultimately prevent the development of depression and anxiety disorders following the onset of insomnia. Research suggests that sleep disruptions lead to emotional dysregulation, including increased negative affectivity and decreased positive affectivity. This affective reactivity may ultimately be related to the development of depression and anxiety. Despite the apparent link between sleep and emotion regulation, studies have not investigated the influence of sleep treatment on these affective dimensions. The investigators long term goal is to increase understanding of the mechanism of action in sleep treatments in relation to changes in positive and negative valence systems. The investigators immediate objective is to conduct a pilot study investigating changes in mean levels and day-to-day instability of affective dimensions following a brief behavioral intervention for insomnia tailored for veterans (Brief Behavioral Treatment for Insomnia-Military Version. The specific aims include developing a deeper understanding of the effects of behavioral sleep treatment on positive and negative valence systems and testing a model in which affective reactivity modulates the relation between sleep and internalizing symptoms. Both objective and subjective sleep data, as well as measures of affective states and depression/anxiety symptoms, will be collected pre and post-treatment in order to examine changes in sleep, affect and daytime symptoms over the course of treatment and to test a model in which affective changes mediate the relation between improvements in sleep and improvements in depression and anxiety. The investigators hypothesize that sleep treatment will improve sleep, daytime symptoms and affective reactivity and that changes in affect will mediate the relation between sleep and internalizing symptoms.

ELIGIBILITY:
Inclusion Criteria:

* meeting Diagnostic and Statistical Manual of Mental Disorders-5 criteria for a diagnosis of insomnia
* a score above the clinical cut-off for insomnia on the Insomnia Severity Index (ISI).63 Participants using psychotropic or hypnotic medications will be eligible if the medication and dose was stable for 3 weeks prior to study entry, and no changes were expected over the course of treatment.

Exclusion Criteria:

* presence of an untreated sleep disorder other than insomnia (e.g., sleep breathing disorder, restless legs syndrome)
* report using drugs or alcohol at high levels
* report moderate or more levels of suicidal or homicidal ideation
* lifetime history of bipolar or psychotic disorder.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | 1 week post-treatment